CLINICAL TRIAL: NCT04717466
Title: Brain Morphological Changes Accompanied by Effective Biologic Treatments for Psoriasis and Their Associations With the Improvement of Well-being, Itch, and Pain
Brief Title: Brain Changes in Psoriasis After Secukinumab Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Gil Yosipovitch, Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20200857
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Psoriasis; Healthy
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Psoriasis Group (Experimental): Psoriasis participants will be given Secukinumab for a total of 4 months. This is a 300mg subcutaneous injection that will occur at weeks 0, 1, 2, 3, 4, 8, and 12.
  Interventions: Biological: Secukinumab
- Healthy Group (No Intervention): Healthy participants will not receive any intervention.

INTERVENTIONS:
Biological: Secukinumab — 300mg subcutaneous injection
  Arms: Psoriasis Group

SUMMARY:
The purpose of this study is to assess the effect of a biologic drug targeting the Interleukin (IL)-17 pathway (secukinumab) on brain plasticity and examine whether the plastic changes correlate with the improvement of perception of well-being, itch, and pain in participants with psoriasis.

ELIGIBILITY:
Inclusion:

1. Between 18 and 65 years of age.
2. Psoriasis patients (with/without psoriatic arthritis): Psoriasis Area (BSA) is more than 5%.
3. Psoriasis patients must have had a TB test in the past 8 months (if a patient has not had one, the study will provide one).
4. Healthy subjects: in general, good health without history of neurological and psychiatric diseases. No chronic itch, pain, skin or systemic conditions currently or in the past.
5. Women of child bearing potential will be administered a pregnancy test to verify that they are not pregnant.
6. MRI Compatibility: No major contraindication for MRI (pacemaker, vascular stents, metallic ear tubes, and absence of metal implants or braces) as assessed by MRI technologist using site approved screening form.
7. Participants have to be able to speak and read English fluently.
8. Participants must have signed a written informed consent before being enrolled in the study

Exclusion:

1. Individuals under 18 or over 65 years of age.
2. Inability to complete the required measures.
3. Participants who use antihistamine drugs for itch relief
4. Suffering from any disease state or physical condition, which would increase their health risk by study participation.
5. Patients with chronic infectious diseases (e.g., mycobacterial and fungal infections and chronic tuberculosis) or inflammatory bowel disease.
6. Patients without a negative TB test in the past 12 months.
7. Hypersensitivity or anaphylaxis to biologics
8. Patients with treatment of biologics should not receive live vaccines. Thus, age appropriate immunizations according to current immunization guidelines must be completed before the experiment.
9. Patients with primary immunodeficient lacking IL-17, patients with autoantibodies against IL-17
10. Currently enrolled in any investigational study in which the subject is receiving any type of drug, biological, or non-drug therapy.
11. Recent initiation (within last 3 months) or change in dose of centrally acting agents such as antidepressants, neuroleptics or neuropathic medications.
12. Patients who were previously treated with drugs targeting IL-17
13. Patients who have used biologics in the past in the past 8 weeks or Otezla in the past 4 weeks.
14. Patients who use centrally acting agents only when they need. The purpose is to avoid a risk of acute effect of these agents on brain activity.
15. Current treatment with opioid analgesics.
16. Uncontrolled thyroid disease.
17. Use of illicit drugs or history of opiate addiction.
18. Diagnosis of a major psychiatric disorder such as schizophrenia, major depression or bipolar disorder that is active currently.
19. Morbid obesity
20. Weight: 250 lb or more
21. Any known diseases or disorders that may affect conducting the experiments (e.g., intracranial pathology, claustrophobia, severe respiratory or cardiovascular problems, active fibromyalgia) or diseases that have potential risks of infections (e.g., HIV, Hepatitis C, etc).
22. Inability to speak and read English.
23. Pregnant.
24. Incarcerated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2025-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gil Yosipovitch, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Psoriasis Group | Healthy Group
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Psoriasis Group | Healthy Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Gray Matter Density
Description: Change in brain anatomy for participants will be reported as the change in average gray matter density as measured by Voxel Based Morphometry (VBM) analysis of Magnetic Resonance Imaging (MRI) scans from baseline to week 4
Time Frame: Baseline to Week 4 (Visit 3)
Measure: Mean (Standard Deviation); unit: voxel
Arm/Group | Psoriasis Group | Healthy Group
Number analyzed (Participants) | 10 | 10
voxel | 0 (0) | 0 (0.000927413)

2. Primary Outcome: Change in Brain Activity
Description: Changes in brain activity in participants will be measured using Arterial Spin Labeling (ASL) MRI from baseline to week 4. ASL quantifies cerebral blood flow CBF in units of ml/100g/min (milliliters of blood per 100 grams of tissue per minute).
Time Frame: Baseline to Week 4 (Visit 3)
Measure: Mean (Standard Deviation); unit: ml/100g/min
Arm/Group | Psoriasis Group | Healthy Group
Number analyzed (Participants) | 10 | 10
ml/100g/min | 1 (55.79089921) | -18 (87.98956788)

3. Secondary Outcome: Change in Itch Score as Measured by the NRS
Description: Itch will be measured using the Numerical Rating Scaling (NRS) ranging from 0 (no itch) to 10 (the worst itch imaginable) baseline to week 4 in psoriasis participant group only.
Time Frame: Baseline to Week 4 (Visit 3)
Population: Only psoriasis patient group included for this analysis as healthy controls were required by enrollment criteria to not have itch.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psoriasis Group
Number analyzed (Participants) | 10
units on a scale | 3 (0.130835626)

4. Secondary Outcome: Change in Pain Score as Measured by the NRS
Description: Pain will be measured using a Numerical Rating Scaling (NRS) ranging from 0 (no pain) to 10 (the worst pain imaginable) baseline to week 4 in psoriasis participant group only.
Time Frame: Baseline to Week 4 (Visit 3)
Population: Only psoriasis patient group included for this analysis as healthy controls were required by enrollment criteria to not have pain.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Psoriasis Group
Number analyzed (Participants) | 10
units on a scale | 2 (0.186739941)

5. Secondary Outcome: Change in PASI Scores
Description: Severity of psoriasis will be measured using the Psoriasis Area and Severity Index (PASI), ranging from 0 to 100 with a higher score indicating more severe psoriasis, from baseline to week 4 in psoriasis participant group only.
Time Frame: Baseline to Week 4 (Visit 3)
Population: Only psoriasis patient group included for this analysis as healthy controls were required by enrollment criteria to not have psoriasis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psoriasis Group
Number analyzed (Participants) | 10
score on a scale | 8 (8.206099453)

6. Secondary Outcome: Change in Participant Well-being as Measured by WHO-5
Description: Well-being will be measured using the 5-item World Health Organization Well-Being Index (WHO-5), ranging from 0 to 25 with a higher score indicating better well-being, from baseline to week 4.
Time Frame: Baseline to Week 4 (Visit 3)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psoriasis Group | Healthy Group
Number analyzed (Participants) | 10 | 10
units on a scale | 2 (0.59336165) | 0 (0.382739698)

7. Secondary Outcome: Change in Quality of Sleep as Measured by a Sleep Numerical Rating Scale Scores
Description: Changes in participants' quality of sleep by using the Numerical Rating Scaling (NRS) ranging from 0 to 10, with a higher score indicating lower sleep quality between baseline, from baseline to week 4.
Time Frame: Baseline to Week 4 (Visit 3)
Population: Initial protocol was to use PSQI survey, but after PI could not get rights for survey use, the protocol was amended to collect sleep disturbance on an NRS scale. Not all study participates completed the Sleep NRS survey, so data was reported on those that did complete this NRS once protocol amendment for its use was IRB approved.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psoriasis Group | Healthy Group
Number analyzed (Participants) | 5 | 7
score on a scale | 0 (0.5) | 2 (1.7)

8. Secondary Outcome: Change in Physical Activity as Measured by 7D-PAR
Description: Physical activity will be measured using the 7-days physical activity recall (7D-PAR), with 0 denoting no exercise and a higher score indicating more physical activity (there is not cap for this score), from baseline to week 4.
Time Frame: Baseline to Week 4 (Visit 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psoriasis Group | Healthy Group
Number analyzed (Participants) | 10 | 10
score on a scale | 7 (9.892384903) | 9 (0.451011454)

9. Secondary Outcome: Changes in Stress in Daily Life as Measured by PSQ
Description: Stress in daily life in psoriasis participants will be measured using the Perceived Stress Questionnaire (PSQ), ranging from 0 to 1 with a higher score indicating more stress, from baseline to week 4.
Time Frame: Baseline, Up to Week 4 (Visit 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psoriasis Group | Healthy Group
Number analyzed (Participants) | 10 | 10
score on a scale | 0.07 (0) | 0.01 (0.01)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Psoriasis Group | Healthy Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psoriasis Group (N=10) | Healthy Group (N=10)
Infected Abcess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Infected Abcess on the left temple
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psoriasis Group (N=10) | Healthy Group (N=10)
itch (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) — itch on the skin or eyes (unrelated or unlikely related to study)
Felt cramped (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient felt cramped for a few second twice on the same day (probably related to study)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Bruising on the skin of the injected site (the right thigh) (related to study)
Swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Swelling of the skin of injected site (left thigh) (related to study)
Nasal and chest congestions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Unrelated to study
tiredness (General disorders) | 1 (2) | 0 (0) — Patient felt tiredness for a couple of day after the initial injection (unrelated to study)
headache (Nervous system disorders) | 1 (1) | 0 (0) — unrelated to study
skin with red/raised/itch (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — On the skin of injected site (both thighs) (related to study)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT04717466/Prot_SAP_000.pdf